CLINICAL TRIAL: NCT02449421
Title: A Comparison of the Effects of Internet-Based Strategies to Support Mental Health Clinicians' Use of an Effective Psychotherapy for Post Traumatic Stress Disorder (PTSD) in Mental Health Systems
Brief Title: Sustaining and Improving Clinicians' Use of Evidence-Based Psychotherapy (EBP) for PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Stanford University (Other); Canadian Institutes of Health Research (CIHR) (Other Government); National Institute of Mental Health (NIMH) (NIH); Palo Alto Veterans Institute for Research (Other); National Center for PTSD (U.S. Federal Agency)
Responsible Party: Principal Investigator, Candice Monson, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB: 2014-345; 137012 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); R01MH106506-01 (NIH)
Record Dates: First submitted 2015-02-09; First posted 2015-05-20 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fidelity-oriented Learning Community (Experimental): The Fidelity-oriented Learning Community arm will receive fidelity consultation (adherence and competence) feedback by a CPT expert via online meetings.
  Interventions: Behavioral: Fidelity-oriented Learning Community
- Quality Improvement Learning Community (Experimental): The Quality Improvement Learning Community arm will include clinicians who set goals related to CPT delivery, execute a plan, study results, refine plan, and continue each cycle until goals are met.
  Interventions: Behavioral: Quality Improvement Learning Community

INTERVENTIONS:
Behavioral: Quality Improvement Learning Community — Consultation with CPT experts to effectively use evidence-based psychotherapy.
  Arms: Quality Improvement Learning Community
Behavioral: Fidelity-oriented Learning Community — The Fidelity-oriented Learning Community arm will receive fidelity consultation (adherence and competence) feedback by a CPT expert via online meetings.
  Arms: Fidelity-oriented Learning Community

SUMMARY:
The purpose of the study is to compare the impact of two strategies to sustain and improve the delivery of an evidence-based psychotherapy for PTSD, Cognitive Processing Therapy (CPT) in three different mental health systems. These approaches are based on two different theories of what is necessary to promote successful implementation. We will examine whether these strategies lead to improved patient outcomes, clinician skill, proportion of clients who receive CPT, and other outcomes that are relevant to the implementation of evidence-based psychosocial treatments. By examining these questions in 3 different mental health systems, we will also examine whether the implementation strategies yield different results in different systems.

DETAILED DESCRIPTION:
This project will compare two different methods of post-training support to promote sustained and improved CPT delivery: Fidelity-oriented learning community (FID-LC) and Continuous Quality Improvement Learning Community (CQI-LC). Clinics in which clinicians have previously received CPT training will be randomly assigned to one of these conditions. Outcomes will be observed changes in patient symptoms during and following treatment, independent expert assessment of clinician fidelity and adaptations in delivering the psychotherapy (via audio-recordings), proportion of eligible caseloads that receive CPT, and capacity to deliver CPT. Data will also be collected to assess clinician and setting characteristics that may contribute to the success of each strategy. The study results will help inform how best to support the ongoing implementation and benefits of evidence-based psychotherapy (e.g., CPT) in routine clinical settings. This is a knowledge translation project in partnership with 3 systems; VA Canada, U.S. Veterans Health Care System and the National Centre for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* All clinicians that provide psychotherapy to patients with PTSD
* Agree to provide CPT to 6 patients over 2 years
* Consent to be randomized to one of two study conditions
* Are willing to record therapy sessions
* Continue to have computer/internet access.
* Patients will be clients of clinician participants that

  1. Are 18 years or older
  2. Have a diagnosis of PTSD
  3. Are willing to have their sessions audiorecorded

Exclusion Criteria:

* Ineligible patient participants are those having

  1. Current uncontrolled psychotic or bipolar disorder
  2. Unremitted substance dependence
  3. Current imminent suicidality or homicidality that requires imminent attention
  4. Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-05-06 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD Symptoms over 6 months (PCL-5 measure) | Participants will be followed for an expected duration of 12 weeks of therapy. PCL-5 will be measured at baseline, at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, post-treatment week, and at 3-month follow-up.
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Each item is measured on a 5-point Likert scale. The PCL will track change from baseline to the 3 month follow up.

SECONDARY OUTCOMES:
Fidelity Measure | At baseline, at 12 and 24 months
  The fidelity measure examines clinicians' adherence and competence to specific CPT interventions prescribed in each session. Clinicians are rated on their adherence to the protocol (on a 0-2 Likert-type scale), as well as their competence in delivery of these elements (rated on a 7-point, Likert-type scale).
Content-Level and Context-Level Adaptation | At baseline, at 12 and 24 months
  Using a framework and coding system of modifications and adaptations made to EBPs, sessions will be rated to identify 11 potential content-level adaptations, as well as 5 context-level modifications.
CPT Activity Reporting | monthly for up to 1 year
  All clinicians will report monthly on CPT activity: caseload size, frequency, duration and satisfaction with the LC over the past month, number of new CPT patients, clinician confidence rating in their CPT delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Candice Monson, PhD, Principal Investigator — Toronto Metropolitan University; Shannon Wiltsey Stirman, PhD, Principal Investigator — National Center for PTSD; Norman Shields, PhD, Principal Investigator — Royal Canadian Mounted Police
Locations (3):
- United States (2):
  - VA Palo Alto Healthcare System, Menlo Park, California
  - UTHSCSA, San Antonio, California
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- [Derived] Thomas FC, Loskot T, Mutschler C, Burdo J, Lagdamen J, Sijercic I, Lane JEM, Liebman RE, Finley EP, Monson CM, Wiltsey-Stirman S. Initiating Cognitive Processing Therapy (CPT) in Community Settings: A Qualitative Investigation of Therapist Decision-Making. Adm Policy Ment Health. 2023 Jan;50(1):137-150. doi: 10.1007/s10488-022-01229-8. Epub 2022 Nov 12. PMID 36370226
- [Derived] Wiltsey Stirman S, Finley EP, Shields N, Cook J, Haine-Schlagel R, Burgess JF Jr, Dimeff L, Koerner K, Suvak M, Gutner CA, Gagnon D, Masina T, Beristianos M, Mallard K, Ramirez V, Monson C. Improving and sustaining delivery of CPT for PTSD in mental health systems: a cluster randomized trial. Implement Sci. 2017 Mar 6;12(1):32. doi: 10.1186/s13012-017-0544-5. PMID 28264720